CLINICAL TRIAL: NCT01958892
Title: To Compare Outcomes After Transurethral Enucleation of Prostate Versus Transurethral Resection of Prostate
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Palaniappan Sundaram, Dr Palaniappan Sundaram, Singapore General Hospital
Other Study IDs: 2012/311/D
Record Dates: First submitted 2013-10-05; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- TURP
  Interventions: Procedure: TURP, TUERP
- TUERP
  Interventions: Procedure: TURP, TUERP

INTERVENTIONS:
Procedure: TURP, TUERP

SUMMARY:
The purpose of the study is to assess whether transurethral enucleation of prostate gives better or equivalent outcomes compared to the gold standard of transurethral resection of the prostate

ELIGIBILITY:
Inclusion Criteria:

* All who underwent TURP or TUERP

Exclusion Criteria:

* Those with prostate cancer, neurogenic bladder, previous urethral or prostate surgery

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: Amles who underwent transurethral prostate surgeryr between 2006 and 2010
Sampling Method: Probability Sample
Dates: Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum urinary flow rate | 6 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - Singapore General Hospital, S'pore, S'pore
  - Singapore General Hospital, Singapore